CLINICAL TRIAL: NCT05565053
Title: Bilateral Erector Spinae Plane Block for Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Halil Cetingok, Ass. Prof, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2019/725
Record Dates: First submitted 2022-08-05; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Myofascial Pain Syndrome
Keywords: Erector spinae plane block; Myofascial pain syndrome; Trigger point; Algometer; Visual Analog Scale; Pain
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain

STUDY DESIGN:
Intervention Model Description: Comparing the efficacy of erector spina plan block and trigger point injection in patients with myofascial pain syndrome
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Erector Spinae Plane Block (Active Comparator): Bilateral Erector Spinae Plane Block
  Interventions: Procedure: Bilateral thoracal erector spinae plane block
- Trigger Point Injection (Active Comparator): Trapezius muscle Trigger Point Injection
  Interventions: Procedure: Trapezius muscle trigger point injection

INTERVENTIONS:
Procedure: Bilateral thoracal erector spinae plane block — Bilateral upper thoracal erector spinae plane block with ultrasound
  Arms: Bilateral Erector Spinae Plane Block
Procedure: Trapezius muscle trigger point injection — Trapezius muscle trigger point injection
  Arms: Trigger Point Injection

SUMMARY:
The investigators aimed to evaluate the effectiveness of bilateral erector spina plane block application in myofascial pain syndrome.

DETAILED DESCRIPTION:
The investigators aimed to evaluate the effectiveness of bilateral erector spina plane block application in myofascial pain syndrome by comparing trigger point injection. Group 1 only one time erector spinae plane block and group 2 once a week total three times trigger point injection. Before the application, one week after application and one month after first application the investigators aimed to compare pressure pain threshold with algometer, visual analog scale score, short form-36 score, neck disability index score, beck depression scale score for the two groups. Each group has 30 participants, total 60 participants included this study. The investigators planned to show that bilateral erector spinae plane block can be used as an effective and safe method in the treatment of myofascial pain syndrome, since it is easier to apply than other invasive procedures used in the treatment and has a very low complication profile.

ELIGIBILITY:
Inclusion Criteria:

* Get a myofascial pain syndrome diagnosis
* No invasive procedure for myofascial pain syndrome in the last 1 month
* Signing the informed consent form

Exclusion Criteria:

* Cervical disc herniation
* Neck/shoulder, thoracal trauma or operation history
* Malignancy
* Kyphoscoliosis
* Inflammatory diseases (Rheumatoid arthritis, ankylosing spondylitis...)
* Congenital vertebral anomalies
* Neck pain with neurological deficit
* Pregnancy
* Mental, psychogenic disorder
* Hematological diseases that cause bleeding and coagulation disorders
* Use of antiplatelet, anticoagulant and drugs that cause bleeding tendency
* Severe systemic infection such as sepsis and local infection at the intervention site
* Having an allergy to any of the drugs to be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-10-27 (Estimated); Study Completion 2022-12-29 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effectiveness of the two interventions (trigger point injection versus Erector spinae plane block) assessed by Visual analog scale (VAS): | Baseline
  The classic interventional treatment of myofascial back pain is trigger point injection. In addition, erector spina plan block has been applied in recent years as an interventional procedure that provides analgesia in the same region and is thought to have a long duration of action. Visual analog scale (VAS): Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Comparison of the effectiveness of the two interventions (trigger point injection versus Erector spinae plane block) assessed by Visual analog scale (VAS): | 1. month
  The classic interventional treatment of myofascial back pain is trigger point injection. In addition, erector spina plan block has been applied in recent years as an interventional procedure that provides analgesia in the same region and is thought to have a long duration of action. Visual analog scale (VAS): Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Çetingök, Study Director — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No